CLINICAL TRIAL: NCT05790733
Title: HYPNONAG : Therapeutic Communication Versus Traditional Method for Naso-gastric Intubation in Haematology: Randomized Controlled Clinical Study
Brief Title: HYPNONAG : Therapeutic Communication Versus Traditional Method for Naso-gastric Intubation in Haematology
Acronym: HYPNONAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC22_9836_HYPNONAG
Record Dates: First submitted 2023-02-13; First posted 2023-03-30 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Aplasia; Chemotherapy Effect
Keywords: Nasogastric intubation
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, bicentric, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (Active Comparator): When the patient is in the conventional arm, the nurse of the service will place the NGS according to the recommendations of the French Health Authorities on the management of the induced pain. The patient is seated at 90 degrees. The nurse takes its landmarks on the NGS to be able to install the NGS at the correct landmark (it takes the NGS and measures "nose-ear, ear-stomach").
  This arm involves the use of the 5% Xylocaine nebulizer spray and a single-use cannula.
  The nurse checks its expiry date and that the quantity is sufficient to practice the 7 instillations in one nostril and the other 7 in the mouth. A waiting time is respected and the installation of the NGS can begin. She will also set up a fast for 2 hours after this local anesthesia.
  Interventions: Other: Standard intubation
- Hypnosis (Experimental): Hypnosis is a particular psychological state marked by the functioning of the individual at a level of attention other than the ordinary state of consciousness. It can, under certain conditions, give the appearance of sleep or somnambulism without sharing all the characteristics.
  As part of the treatment, hypnosis is widely used for pain control. The adverse effects reported are nil. One of its main benefits is improved patient comfort. Another benefit is the reduction of exposure to anesthetic products.
  The installation of the SNG with hypnosis will be carried out according to the protocol set out in appendix 4.
  In the hypnosis arm, there will be none local anesthesia.
  Interventions: Other: Hypnosis

INTERVENTIONS:
Other: Standard intubation — This involves the use of 5% Xylocaine nebulizer spray and a single-use cannula. The nurse checks its expiry date and that the quantity is sufficient to practice the 7 instillations in one nostril and the other 7 in the mouth. A waiting time is respected and the installation of the NGS can begin. She will also set up a fast for 2 hours after this local anesthesia.
  Arms: Standard
Other: Hypnosis — Hypnosis is a particular psychological state marked by the functioning of the individual at a level of attention other than the ordinary state of consciousness. It can, under certain conditions, give the appearance of sleep or somnambulism without sharing all the characteristics.
  As part of the treatment, hypnosis is widely used for pain control. The adverse effects reported are nil. One of its main benefits is improved patient comfort. Another benefit is the reduction of exposure to anesthetic products.
  The installation of the NGS with hypnosis will be carried out according to the protocol set out in appendix 4.
  Arms: Hypnosis

SUMMARY:
Caloric intake is a determining factor in patients with hematological malignancies and hospitalized for prolonged aplasia following chemotherapy. The nutritional supplement is administered either parenterally or enterally through the placement of a nasogastric sonde (NGS). This last option has shown its advantage compared to parenteral nutrition in terms of preventing infections, the incidence of graft-versus-host disease in allograft patients, and the quality of resumption of oral nutrition during of returning home.

NGS allows the administration of an intake of 2000 calories/day, deemed necessary to mitigate the risk of undernutrition in patients hospitalized for more than 3 weeks and in the majority of cases unable to eat enough food mainly due to chemotherapy-induced mucositis. . The choice between enteral feeding by NGS and parenteral nutrition is the subject of controversial studies, with each team choosing one of the two options.

The installation of the NGS is often recognized as a traumatic gesture for patients but also invasive by caregivers.

The patient's anxiety, the intrusive and traumatic nature of the NGS can sometimes result in a failure of the gesture, a secondary refusal of the patient, or a reluctance of the caregiver to proceed with the gesture. Since 2013, NGS have been placed with the assistance of the nurse who practices hypnosis in the hematology department of the Rennes University Hospital. This invites the patient to pose his SNG without local anesthesia and in a completely autonomous way. The patient is thus able to place the NGS again if necessary during his hospitalization, and during subsequent hospitalizations. A retrospective and monocentric study carried out at the University Hospital of Rennes in 38 patients showed that all were able to perform NGS independently thanks to the hypnotic approach. It was observed a real comfort for the patient, and moreover this technique did not add extra work for the staff. The patient becomes autonomous and actor of his care.

DETAILED DESCRIPTION:
Strategy : Hypnosis versus standard way for the installation of an NGS. In the conventional arm, the nurse will place the NGS according to the recommendations of the French Health Authorities on the management of the induced pain. The patient is seated at 90 degrees. The nurse takes its landmarks on the NGS to be able to install the NGS at the correct landmark (it takes the SNG and measures "nose-ear, ear-stomach").

As part of this project, local anesthesia will be performed if the patient is part of the control arm and there will be none if he is part of the hypnosis arm.

When the patient will be randomized in the hypnosis arm, he will place his NGS himself with a hypnotic accompaniment, described in appendix.

This original project aims to evaluate the contribution of hypnosis in the installation of an NGS in patients hospitalized for the management of a malignant hemopathy for a period of at least 3 weeks. A group of patients will benefit from the autonomous installation of the NGS thanks to the assistance of a nurse hypnotherapist and will be compared to a group of patients for whom the NGS will be set up in a standard way. The main expected benefits of hypnosis for the patient include improved comfort and near absence of discomfort or pain during NGS placement, minimal anxiety and ultimately a benefit in terms of caloric intake administered during prolonged hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for chemotherapy generating an aplasia lasting more than 8 days (hospitalization for 3 weeks) and for whom the insertion of an NGS is required and not yet attempted since admission to the hospital;
* Age ≥ 18 years;
* Affiliated to a social security scheme;
* Having signed a free, informed and written consent.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Patient who refuses NGS;
* Emergency surgery;
* Patients consuming long-term opiates before surgery;
* Substance addiction;
* Patient at the end of life and/or in palliative care;
* Patient unable to answer a questionnaire and/or unable to understand the rating scales;
* Deaf and/or dumb patients;
* Patients with psychiatric pathologies (schizophrenia, bipolarity);
* Persons subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Comfort | Within 3 minutes after the end of the intubation
  Patient comfort will be assessed by a simple, validated digital comfort scale. This scale is graduated from "0" (no comfort) to "10" (maximum conceivable comfort). This evaluation will be carried within 3 minutes following the end of the intubation, i.e. after having checked the correct location of the probe thanks to the presence of air blown in by a syringe with a conical tip, that the nurse will check with a stethoscope right after securing the SNG with a hypoallergenic dressing on the patient's chee

SECONDARY OUTCOMES:
Pain visual analogue scale | Immediately after the assessment of the comfort scale (assessed within 3 minutes after the end of the intubation)
  The patient's pain will be assessed by the visual analogue scale (VAS). This scale is graduated from "0" (no pain) to "10" (maximum pain imaginable). It will be performed immediately after the assessment of the comfort scale.
Anxiety | 5 minutes (+/- 1 minute) before the NGS placement starts and repeated immediately after the procedure ends (just after the pain assessment)
  The anxiety felt by the patient will be assessed by a simple and validated numerical scale. This scale is graduated from "0" (no anxiety) to "10" (maximum anxiety imaginable). It will be performed 10 minutes (+/- 3 minutes) before the biopsy procedure and repeated after the biopsy procedure (just after the pain assessment).
Success or failure of the NGS placement according to the randomization arm | During procedure
  Success or failure of the NGS placement after using the method (standard method versus hypnosis) given by the randomization arm
Number of failures | During procedure
  The number of failures during the first NGS insertion according to the randomization arm with the need to switch to another NGS insertion procedure, or even the need to switch to parenteral nutrition (following repeated failures of the NGS).
Weight | From date of admission to hospital in the hematology department up to date of the hospital discharge in the hematology department, assessed up to 3 months
  Weight at entry and exit from hospitalization in the hematology department.
Muscular strength | From date of admission to hospital in the hematology department up to date of the hospital discharge in the hematology department, assessed up to 3 months
  Muscular strength assessed by means of a dynamometer at entry and exit from hospitalization in the hematology department
Total number of days of presence of the NGS | During the hospitalization time (up to 3 months)
  The total number of days of presence of the NGS during the hospitalization time
Attempt or not of a new NGS intubation (in case of rejection of the first probe by vomiting) | From date of admission to hospital in the hematology department up to date of the hospital discharge in the hematology department, assessed up to 3 months
  In case of rejection of the first probe by vomiting during hospitalization, attempt or not of a new NGS intubation

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Rennes University Hospital, Rennes, Brittany Region
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No